CLINICAL TRIAL: NCT00885313
Title: Study of Efficacy and Tolerability of Docosahexaenoic Acid (DHA) on Children Affected by Nonalcoholic Fatty Liver Disease (NAFLD).
Brief Title: Effects of Docosahexaenoic Acid (DHA) on Children With Nonalcoholic Fatty Liver Disease (NAFLD)
Acronym: EDACN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Valerio Nobili, MD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1406-18-4
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Fatty Liver; Liver Fibrosis; Obesity; Metabolic Syndrome; Nonalcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; fibrosis
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Obesity; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — Docosahexaenoic Acids; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DHA250 (Experimental): DHA 250 mg/kg/d plus lifestyle intervention [hypocaloric Diet (25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Interventions: Drug: DHA250; Behavioral: Lifestyle intervention
- DHA500 (Experimental): DHA 250 mg/kg/d plus lifestyle intervention [hypocaloric Diet (25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Interventions: Drug: DHA500; Behavioral: Lifestyle intervention
- PLA (Placebo Comparator): placebo and lifestyle intervention [hypocaloric Diet (25-30 cal/kg/d) or isocaloric (40-45 cal/kg/d) and physical activity].
  Interventions: Drug: PLACEBO; Behavioral: Lifestyle intervention

INTERVENTIONS:
Drug: DHA250 — DHA 250 mg/kg/d
  Other Names: Docosahexaenoic Acid
  Arms: DHA250
Drug: DHA500 — DHA 500 mg/kg/d
  Other Names: Docosahexaenoic Acid
  Arms: DHA500
Drug: PLACEBO — placebo
  Other Names: No interventions
  Arms: PLA
Behavioral: Lifestyle intervention — lifestyle intervention [including hypocaloric diet (25-30 cal/kg/d) or isocaloric diet (40-45 cal/kg/d) and physical activity], for 12 months.
  Other Names: Diet and physical activity

SUMMARY:
The purpose of this interventional study is to evaluate the efficacy and tolerability of docosahexaenoic acid (DHA) in children or adolescents with well-characterized and liver biopsy confirmed nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Sixty children or adolescents (4-16 years) with liver biopsy proven NAFLD will be enrolled. They will be randomized to treatment with DHA 250 mg/kg/d (n=20), DHA 500 mg/kg/d (n=20), or an identical placebo (n=20) given orally for a period of 24 months. All patients will be included in a lifestyle intervention program consisting of a diet tailored on the individual requirements and physical exercise.

Patients will undergo a medical evaluation every three months during the 24-month study period. Liver biopsy will be performed only at baseline and at the end of treatment. Anthropometric analysis, laboratory tests, including liver enzymes and lipids will be repeated at 3-month intervals during the 24-month study duration. Ultrasonography and Fibroscan of the liver will be repeated at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* persistently elevated serum aminotransferase levels
* diffusely echogenic liver on imaging studies suggestive of fatty liver
* biopsy consistent with the diagnosis of NAFLD

Exclusion Criteria:

* hepatic virus infections (HCV RNA-PCR negative)
* Hepatitis A, B, C, D, E and G
* cytomegalovirus and Epstein-Barr virus
* alcohol consumption
* history of parenteral nutrition
* use of drugs known to induce steatosis or to affect body weight and carbohydrate metabolism
* autoimmune liver disease, metabolic liver disease, Wilson's disease, and a-1-antitrypsin-associated liver disease were ruled out using standard clinical, laboratory and histological criteria

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Liver status by liver biopsy (steatosis and fibrosis) | months 24

SECONDARY OUTCOMES:
Serum alanine transferase levels | month 24
Serum levels of triglycerides | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, MD, Principal Investigator — Bambino Gesù Children Hospital
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Rome, Italy

REFERENCES:
- [Derived] Nobili V, Bedogni G, Donati B, Alisi A, Valenti L. The I148M variant of PNPLA3 reduces the response to docosahexaenoic acid in children with non-alcoholic fatty liver disease. J Med Food. 2013 Oct;16(10):957-60. doi: 10.1089/jmf.2013.0043. Epub 2013 Sep 28. PMID 24074360
- [Derived] Nobili V, Alisi A, Della Corte C, Rise P, Galli C, Agostoni C, Bedogni G. Docosahexaenoic acid for the treatment of fatty liver: randomised controlled trial in children. Nutr Metab Cardiovasc Dis. 2013 Nov;23(11):1066-70. doi: 10.1016/j.numecd.2012.10.010. Epub 2012 Dec 7. PMID 23220074
- [Derived] Nobili V, Bedogni G, Alisi A, Pietrobattista A, Rise P, Galli C, Agostoni C. Docosahexaenoic acid supplementation decreases liver fat content in children with non-alcoholic fatty liver disease: double-blind randomised controlled clinical trial. Arch Dis Child. 2011 Apr;96(4):350-3. doi: 10.1136/adc.2010.192401. Epub 2011 Jan 12. PMID 21233083